CLINICAL TRIAL: NCT00496197
Title: Phase IV Open Label Non Comparative Trial Of IV Anidulafungin Followed By Oral Azole Therapy For The Treatment Of Candidemia And Invasive Candidiasis
Brief Title: Study Will Evaluate The Safety And Efficacy Of Anidulafungin In Patients With Candidemia Or Invasive Candidiasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8851011
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Candidiasis
Keywords: candidemia; invasive candidiasis; fungal bloodstream infection
MeSH Terms: conditions — Candidiasis; Candidemia; Candidiasis, Invasive | interventions — Anidulafungin; Fluconazole; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1. (Experimental): Subjects receive anidulafungin IV followed by oral therapy with fluconazole or voriconazole.
  Interventions: Drug: Eraxis (anidulafungin); Drug: Diflucan (fluconazole); Drug: Vfend (voriconazole)

INTERVENTIONS:
Drug: Eraxis (anidulafungin) — Subjects will receive IV anidulafungin (200 mg loading dose followed by 100 mg maintenance doses QD) for 5-28 days. This will be followed by oral therapy with fluconazole at 400 mg once daily or voriconazole at 200 mg twice daily until 14 days after the last positive culture. Fluconazole will be used if the baseline cultures are positive for C. albicans or C. parapsilosis while voriconazole will be used if cultures are positive for C. glabrata or other non-albicans species.
Drug: Diflucan (fluconazole) — Subjects will receive IV anidulafungin (200 mg loading dose followed by 100 mg maintenance doses QD) for 5-28 days. This will be followed by oral therapy with fluconazole at 400 mg once daily or voriconazole at 200 mg twice daily until 14 days after the last positive culture. Fluconazole will be used if the baseline cultures are positive for C. albicans or C. parapsilosis.
Drug: Vfend (voriconazole) — Subjects will receive IV anidulafungin (200 mg loading dose followed by 100 mg maintenance doses QD) for 5-28 days. This will be followed by oral therapy with fluconazole at 400 mg once daily or voriconazole at 200 mg twice daily until 14 days after the last positive culture. Fluconazole will be used if the baseline cultures are positive for C. albicans or C. parapsilosis while voriconazole will be used if cultures are positive for C. glabrata or other non-albicans species.

SUMMARY:
The purpose of this study is to further evaluate the safety and effectiveness of intravenous anidulafungin (Eraxis™) in patients with a diagnosis of candidemia or invasive candidiasis, which is a fungus infection of the blood or tissue. Currently the drug is approved for treatment using a daily dose of IV medication until 14 days after the fungus disappears from the blood. This study will evaluate the effectiveness of intravenous anidulafungin when it is administered for 5-28 days followed by oral antifungal medication. Study patients will be assessed for response to treatment throughout the study drug treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > or equal to 18 years of age.
* Presence of candidemia (positive blood culture) or invasive candidiasis (histopathologic or cytopathologic examination of a needle aspiration or biopsy specimen from a normally sterile site excluding mucous membranes showing yeast cells) obtained within the prior 96 hours of the screening visit.
* Subjects who received no more than one prior dose of an echinocandin or polyene.

Exclusion Criteria:

* Subjects with hypersensitivity to anidulafungin, other echinocandins or azoles.
* Presence of confirmed or suspected Candida osteomyelitis, endocarditis or meningitis.
* Subjects with infected prosthetic devices which cannot be removed within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (29):
- United States (28):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Minneota, Minnesota
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Camden, New Jersey
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Houston, Texas
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- [Derived] De Rosa FG, Busca A, Capparella MR, Yan JL, Aram JA. Invasive Candidiasis in Patients with Solid Tumors Treated with Anidulafungin: A Post Hoc Analysis of Efficacy and Safety of Six Pooled Studies. Clin Drug Investig. 2021 Jun;41(6):539-548. doi: 10.1007/s40261-021-01024-7. Epub 2021 Apr 23. PMID 33891293
- [Derived] Sganga G, Wang M, Capparella MR, Tawadrous M, Yan JL, Aram JA, Montravers P. Evaluation of anidulafungin in the treatment of intra-abdominal candidiasis: a pooled analysis of patient-level data from 5 prospective studies. Eur J Clin Microbiol Infect Dis. 2019 Oct;38(10):1849-1856. doi: 10.1007/s10096-019-03617-9. Epub 2019 Jul 6. PMID 31280481
- [Derived] Kontoyiannis DP, Bassetti M, Nucci M, Capparella MR, Yan JL, Aram J, Hogan PA. Anidulafungin for the treatment of candidaemia caused by Candida parapsilosis: Analysis of pooled data from six prospective clinical studies. Mycoses. 2017 Oct;60(10):663-667. doi: 10.1111/myc.12641. Epub 2017 Jun 9. PMID 28597967
- [Derived] Kullberg BJ, Vasquez J, Mootsikapun P, Nucci M, Paiva JA, Garbino J, Yan JL, Aram J, Capparella MR, Conte U, Schlamm H, Swanson R, Herbrecht R. Efficacy of anidulafungin in 539 patients with invasive candidiasis: a patient-level pooled analysis of six clinical trials. J Antimicrob Chemother. 2017 Aug 1;72(8):2368-2377. doi: 10.1093/jac/dkx116. PMID 28459966
- [Derived] Vazquez J, Reboli AC, Pappas PG, Patterson TF, Reinhardt J, Chin-Hong P, Tobin E, Kett DH, Biswas P, Swanson R. Evaluation of an early step-down strategy from intravenous anidulafungin to oral azole therapy for the treatment of candidemia and other forms of invasive candidiasis: results from an open-label trial. BMC Infect Dis. 2014 Feb 21;14:97. doi: 10.1186/1471-2334-14-97. PMID 24559321
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851011&StudyName=Study%20Will%20Evaluate%20The%20Safety%20And%20Efficacy%20Of%20Anidulafungin%20In%20Patients%20With%20Candidemia%20Or%20Invasive%20Candidiasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin: Anidulafungin 200 milligrams (mg) intravenous (IV) loading dose followed by 100 mg IV infusion once a day (QD) for a minimum of 5 days and up to a maximum of 28 days. Participants who complete a minimum of 5 days IV treatment may be switched to oral (PO) fluconazole or voriconazole therapy any day between Day 6 and 28 dependent on criteria that includes negative blood cultures. Participants will continue on antifungal treatment for a minimum of 14 days after last positive blood and / or tissue culture and resolution of signs and symptoms of fungal infection.
Period: Overall Study
Arm/Group | Anidulafungin
Started | 282
Completed | 160
Not Completed | 122
Not completed — Discontinued study due to death | 43
Not completed — Adverse Event | 13
Not completed — Does not meet entrance criteria | 5
Not completed — Insufficient clinical response | 3
Not completed — Insufficient bacteriological response | 10
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 11
Not completed — Pathogen not isolated baseline specimen | 4
Not completed — Other | 14
Not completed — Protocol Violation | 8

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin
Number analyzed (Participants) | 282
Age, Customized [Number; unit: participants]
  18 to 44 years of age | 72
  45 to 64 years of age | 116
  ≥ 65 years of age | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131
  Male | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Global Response of Success or Failure (Based on Clinical and Microbiological Response) at End of Treatment (EOT)
Description: Success: Clinical response=Cure (no signs, symptoms [s/s] of Candida) or Improvement (significant, incomplete resolution of s/s) and Microbiological response=Eradication (follow up [f/u] culture negative) or Presumed Eradication (f/u culture not available [n/a] and response of clinical success). Failure: Clinical response=Failure (≥3 doses Anidulafungin with no significant improvement in s/s or death due to Candida) and Microbiological response=Persistence (positive culture for ≥1 baseline Candida species [spp]) or Presumed Persistence (f/u culture n/a and clinical outcome= failure).
Time Frame: End of Treatment (Day 5 up to Day 42)
Population: Modified Intent to Treat population (MITT): includes all participants who received at least 1 dose of study medication and with a positive baseline culture for a Candida spp. N=number of participants included in analysis (participants with missing outcome values were excluded from the analysis).
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 203
participants
  Success (Cure or Improvement) | 170
  Failure | 33
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at EOT; Test type: Superiority or Other; percentage of participants = 83.7, 95% CI 2-sided [78.7 to 88.8] — 95% Confidence interval based on normal approximation to the binomial. Percentages based on the number of participants in analysis

2. Secondary Outcome: Number of Participants With Clinical Response at EOT
Description: Clinical Success=Cure: resolution of Candida s/s or Improvement: significant but incomplete resolution of s/s; Clinical Failure: at least 3 doses Anidulafungin with no significant improvement in s/s or death due to Candida.
Time Frame: End of Treatment (Day 5 up to Day 42)
Population: MITT; N=number of participants included in analysis (participants with missing outcome values were excluded from the analysis).
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 187
participants
  Cure | 160
  Improvement | 14
  Failure | 13
Statistical Analysis 1: Comparison: Anidulafungin; Clinical response of Success (cure or improvement) at EOT; Test type: Superiority or Other; percentage of participants = 93.0, 95% CI 2-sided [89.4 to 96.7] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Microbiological Response at EOT
Description: Microbiological Success=Eradication: negative culture for baseline Candida spp or Presumed Eradication: f/u culture n/a and clinical outcome defined as success (cure or improvement); Microbiological Failure=Persistence: positive culture for at least 1 baseline Candida spp or Presumed Persistence: f/u culture n/a and clinical outcome defined as failure (≥3 doses Anidulafungin with no significant improvement in s/s or death due to Candida).
Time Frame: End of Treatment (Day 5 up to Day 42)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 192
participants
  Eradication | 124
  Presumed eradication | 59
  Persistence | 6
  Presumed persistence | 3
Statistical Analysis 1: Comparison: Anidulafungin; Microbiological response of Success (eradication or presumed eradication) at EOT; Test type: Superiority or Other; percentage of participants = 95.3, 95% CI 2-sided [92.3 to 98.3] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Global Response of Success or Failure (Based on Clinical and Microbiological Response) at End of Intravenous Treatment (EOIV)
Description: Success: Clinical response=Cure (s/s of Candida) or Improvement (significant, incomplete resolution of s/s) and Microbiological response=Eradication (f/u culture negative) or Presumed Eradication (f/u culture n/a and response of clinical success). Failure: Clinical response=Failure (≥3 doses Anidulafungin with no significant improvement in s/s or death due to Candida) and Microbiological response=Persistence (positive culture for ≥1 baseline Candida spp) or Presumed Persistence (f/u culture n/a and clinical outcome= failure).
Time Frame: End of Intravenous treatment (Day 5 up to Day 28)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 235
participants
  Success (Cure or Improvement) | 208
  Failure | 27
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at EOIV; Test type: Superiority or Other; percentage of participants = 88.5, 95% CI 2-sided [84.4 to 92.6] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Clinical Response at EOIV
Description: as for outcome 2
Time Frame: End of Intravenous treatment (Day 5 up to Day 28)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 232
participants
  Cure | 159
  Improvement | 57
  Failure | 16
Statistical Analysis 1: Comparison: Anidulafungin; Clinical response of Success (cure or improvement) at EOIV; Test type: Superiority or Other; percentage of participants = 93.1, 95% CI 2-sided [89.8 to 96.4] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With Microbiological Response at EOIV
Description: as for outcome 3
Time Frame: End of Intravenous treatment (Day 5 up to Day 28)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 242
participants
  Eradication | 163
  Presumed eradication | 61
  Persistence | 15
  Presumed persistence | 3
Statistical Analysis 1: Comparison: Anidulafungin; Microbiological response of Success (eradication or presumed eradication) at EOIV; Test type: Superiority or Other; percentage of participants = 92.6, 95% CI 2-sided [89.3 to 95.9] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Sustained (Continued) Global Response of Success or Failure (Based on Clinical and Microbiological Response) at Week 2 Follow-up
Description: as for outcome 4
Time Frame: Week 2 Follow-up
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 194
participants
  Success (Cure or Improvement) | 148
  Failure | 46
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at Week 2 Follow-up; Test type: Superiority or Other; percentage of participants = 76.3, 95% CI 2-sided [70.3 to 82.3] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Number of Participants With Sustained (Continued) Clinical Response at Week 2 Follow-up
Description: as for outcome 2
Time Frame: Week 2 follow-up
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 173
participants
  Cure | 155
  Improvement | 9
  Failure | 9
Statistical Analysis 1: Comparison: Anidulafungin; Clinical response of Success (cure or improvement) at Week 2 Follow-up; Test type: Superiority or Other; percentage of participants = 94.8, 95% CI 2-sided [91.5 to 98.1] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Number of Participants With Sustained (Continued) Microbiological Response at Week 2 Follow-up
Description: as for outcome 3
Time Frame: Week 2 Follow-up
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 173
participants
  Eradication | 30
  Presumed eradication | 135
  Persistence | 3
  Presumed persistence | 5
Statistical Analysis 1: Comparison: Anidulafungin; Microbiological response of Success (eradication or presumed eradication) at Week 2 Follow-up; Test type: Superiority or Other; percentage of participants = 95.4, 95% CI 2-sided [92.2 to 98.5] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Number of Participants With Sustained (Continued) Global Response of Success or Failure (Based on Clinical and Microbiological Response) at Week 6 Follow-up (End of Study [EOS])
Description: as for outcome 4
Time Frame: Week 6 Follow-up (EOS)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 187
participants
  Success (Cure or Improvement) | 131
  Failure | 56
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at Week 6 Follow-up (EOS); Test type: Superiority or Other; percentage of participants = 70.1, 95% CI 2-sided [63.5 to 76.6] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Participants With Sustained (Continued) Clinical Response at Week 6 Follow-up (EOS)
Description: as for outcome 2
Time Frame: Week 6 follow-up (EOS)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 156
participants
  Cure | 138
  Improvement | 8
  Failure | 10
Statistical Analysis 1: Comparison: Anidulafungin; Clinical response of Success (cure or improvement) at Week 6 Follow-up (EOS); Test type: Superiority or Other; percentage of participants = 93.6, 95% CI 2-sided [89.7 to 97.4] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Number of Participants With Sustained (Continued) Microbiological Response at Week 6 Follow-up (EOS)
Description: as for outcome 3
Time Frame: Week 6 Follow-up (EOS)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 156
participants
  Eradication | 12
  Presumed eradication | 134
  Persistence | 2
  Presumed persistence | 8
Statistical Analysis 1: Comparison: Anidulafungin; Microbiological response of Success (eradication or presumed eradication) at Week 6 Follow-up (EOS); Test type: Superiority or Other; percentage of participants = 93.6, 95% CI 2-sided [89.7 to 97.4] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Number of Participants With Global Response of Success or Failure (Based on Clinical and Microbiological Response) at EOT for Participants With Non-albicans Candida at Baseline
Description: as for outcome 4
Time Frame: End of Treatment (Day 5 up to Day 42)
Population: MITT; N=number of participants in the MITT population where the pathogen isolated at baseline was a Candida spp. other than Candida albicans (participants with missing outcome values were excluded from the analysis).
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 120
participants
  Success (Cure or Improvement) | 99
  Failure | 21
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at EOT; Test type: Superiority or Other; percentage of participants = 82.5, 95% CI 2-sided [75.7 to 89.3] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Number of Participants With Global Response of Success or Failure (Based on Clinical and Microbiological Response) at EOIV for Participants With Non-albicans Candida at Baseline
Description: as for outcome 4
Time Frame: End of Intravenous treatment (Day 5 up to Day 28)
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 139
participants
  Success (Cure or Improvement) | 119
  Failure | 20
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at EOIV; Test type: Superiority or Other; percentage of participants = 85.6, 95% CI 2-sided [79.8 to 91.4] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Number of Participants With Global Response of Success or Failure (Based on Clinical and Microbiological Response) at Week 2 Follow-up for Participants With Non-albicans Candida at Baseline
Description: as for outcome 4
Time Frame: Week 2 Follow-up
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 116
participants
  Success (Cure or Improvement) | 89
  Failure | 27
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at Week 2 Follow-up; Test type: Superiority or Other; percentage of participants = 76.7, 95% CI 2-sided [69.0 to 84.4] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Number of Participants With Global Response of Success or Failure (Based on Clinical and Microbiological Response) at Week 6 Follow-up (EOS) for Participants With Non-albicans Candida at Baseline
Description: as for outcome 4
Time Frame: Week 6 Follow-up (EOS)
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 111
participants
  Success (Cure or Improvement) | 75
  Failure | 36
Statistical Analysis 1: Comparison: Anidulafungin; Global response of Success (cure or improvement) at Week 6 Follow-up (EOS); Test type: Superiority or Other; percentage of participants = 67.6, 95% CI 2-sided [58.9 to 76.3] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Time (75% Quartile Point Estimate) to Negative Blood and / or Tissue Culture for Candida Species
Description: Participants with a negative culture on Day 1 were not included in the analysis. For participants with a positive culture on Day 1, the first day on which there was a negative culture was determined and then compared to the result of the next culture. If the next culture was also negative, or the next culture was positive but the interval between the 2 cultures was > 3 days, the earlier of the 2 cultures was the day of first negative blood culture. If next culture was positive and taken within 3 days of the previous culture, the process was repeated with the next negative blood culture.
Time Frame: Baseline (Day 1) up to Week 6 Follow-up (EOS)
Population: MITT; Confidence interval (CI) for the median could not be calculated by the software because no event time met the criteria for inclusion into the CI.
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 282
days | 3.0000 [2.0000 to 3.0000]

18. Secondary Outcome: Medical Resource Utilization (MRU): Duration of Hospital Stay (Days)
Description: Measured as time to dischargeable (medically dischargeable status) and as time to discharge (actual discharge). Analysis of length of hospital stay based on Kaplan-Meier survival techniques.
Time Frame: Baseline up to 6 Week Follow-up (EOS)
Population: MITT; N=number of participants with analyzable data at observation. Time to dischargeable and time to discharge censored at Week 6 Follow-up (EOS).
Measure: Mean (Standard Error); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 248
days
  Time to dischargeable | 27.3 (3.24)
  Time to discharge | 27.1 (3.02)

19. Secondary Outcome: Medical Resource Utilization (MRU): Duration of Intensive Care Unit or Critical Care Unit Stay (Days)
Description: Analysis of length of hospital stay based on Kaplan-Meier survival techniques.
Time Frame: Baseline up to 6 Week Follow-up (EOS)
Population: MITT; N=number of participants with analyzable data at observation. Length of hospital stay censored at Week 6 Follow-up (EOS).
Measure: Mean (Standard Error); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 108
days | 18.4 (2.11)

20. Secondary Outcome: Medical Resource Utilization (MRU): Duration of Intravenous Therapy (Days)
Description: Analysis of length of hospital stay based on Kaplan-Meier survival techniques.
Time Frame: Baseline up to End of Intravenous treatment (Day 5 up to Day 28)
Population: as for outcome 19
Measure: Mean (Standard Error); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 250
days | 8.9 (0.37)

21. Secondary Outcome: Medical Resource Utilization (MRU): Duration of Overall Therapy (Days)
Description: Overall therapy includes Intravenous and Oral therapy. Participants were to receive at least 5 days and a maximum of 28 days of IV anidulafungin. After that, participants could continue treatment with oral fluconazole or voriconazole for at least 14 days from the day of last positive culture.
Time Frame: Baseline up to End of Treatment (Day 5 up to Day 42)
Population: Intent to Treat (ITT) population includes all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 282
days | 14.1 (8.21)

22. Secondary Outcome: Number of Participants Per Specified Cause of Death
Description: Cause of death (includes all-cause and attributable to Candida infection) reported based on death due to Serious Adverse Events (SAEs). SAEs are any untoward medical occurrence at any dose that results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, results in congenital anomaly or birth defect. Participants may be counted with > 1 cause of death if multiple causes were present.
Time Frame: Baseline up to Week 6 Follow-up (EOS) or 30 days after last dose of study drug (whichever was later)
Population: Safety analysis set is the same as the Intent-to-Treat population (ITT) and includes all participants who had taken at least 1 dose of study medication. N=number of participants who died with cause of death reported as Serious Adverse Events.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 65
participants
  Acute myocardial infarction | 1
  Acute respiratory failure | 1
  Anastomotic complication | 1
  Ascites | 2
  Atrial flutter | 1
  Bile duct cancer | 1
  Brain oedema | 1
  Cardiac arrest | 5
  Cardiac failure congestive | 1
  Cardio-respiratory arrest | 1
  Chronic hepatic failure | 2
  Coagulopathy | 1
  Colon cancer | 1
  Convulsion | 1
  Deep vein thrombosis | 1
  Diabetes mellitus | 1
  Disease progression | 8
  Dyspnoea | 1
  Electromechanical dissociation | 1
  Endocarditis | 1
  Endotracheal intubation | 1
  Fungaemia | 1
  Gastrointestinal haemorrhage | 1
  Gastrointestinal ischaemia | 1
  General physical health deterioration | 1
  Haemorrhage | 1
  Haemorrhage intracranial | 1
  Hepatic failure | 1
  Hypoglycaemia | 2
  Hyponatraemia | 1
  Hypotension | 2
  Infection | 1
  Ischaemic cardiomyopathy | 1
  Liver function test abnormal | 1
  Lymphoma | 3
  Mental status changes | 1
  Metastatic gastric cancer | 1
  Multi-organ disorder | 1
  Multi-organ failure | 4
  Multiple myeloma | 1
  Multiple sclerosis relapse | 1
  Myocardial infarction | 1
  Neoplasm malignant | 1
  Peritonitis | 1
  Peritonitis bacterial | 1
  Pneumonia | 3
  Pneumothorax | 1
  Pulmonary embolism | 1
  Pulmonary haemorrhage | 1
  Renal failure | 5
  Renal failure acute | 1
  Renal failure chronic | 1
  Respiratory arrest | 3
  Respiratory distress | 2
  Respiratory failure | 6
  Sepsis | 12
  Septic shock | 7
  Systemic candida | 1
  Thrombocytopenia | 1
  Wound dehiscence | 1

23. Secondary Outcome: Number of Participants With Non-serious and Serious Adverse Events
Description: AEs are any untoward medical occurrence in a clinical investigation subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. SAEs are any untoward medical occurrence at any dose that results in death, is life threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, results in congenital anomaly or birth defect.
Time Frame: Baseline up to Week 6 Follow-up (EOS) or 30 days after last dose of study drug (whichever was later)
Population: Safety analysis set. An event may have been reported as both a serious and non-serious adverse event, however, what is presented are distinct events; participants may be counted as having experienced > 1 event.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 282
participants
  Non-serious Adverse Events | 216
  Serious Adverse Events | 134

24. Secondary Outcome: Number of Participants Who Died
Time Frame: Baseline up to Week 6 Follow-up (EOS) or 30 days after last dose of study drug (whichever was later)
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 282
participants | 65

ADVERSE EVENTS:
Time Frame: Baseline up to Week 6 Follow-up (EOS)or 30 days after last dose of study drug (whichever was later)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Anidulafungin
Serious Adverse Events (participants affected / at risk) | 134/282
Other Adverse Events (participants affected / at risk) | 132/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=282)
Coagulopathy (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 6
Cardiac failure (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Electromechanical dissociation (Cardiac disorders) | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Mitral valve disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Pancreatitis acute (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Device malfunction (General disorders) | 1
Disease progression (General disorders) | 5
Local swelling (General disorders) | 1
Multi-organ disorder (General disorders) | 1
Multi-organ failure (General disorders) | 4
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Chronic hepatic failure (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Abdominal abscess (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 4
Bacterial sepsis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 4
Cytomegalovirus infection (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Fungal endocarditis (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Pancreatic abscess (Infections and infestations) | 1
Pelvic abscess (Infections and infestations) | 1
Peridiverticular abscess (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pseudomembranous colitis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 13
Septic shock (Infections and infestations) | 9
Systemic candida (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection bacterial (Infections and infestations) | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Bleeding time prolonged (Investigations) | 1
Blood culture positive (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anoxic encephalopathy (Nervous system disorders) | 1
Brain oedema (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Haemorrhage intracranial (Nervous system disorders) | 1
Intracranial hypotension (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 4
Renal failure (Renal and urinary disorders) | 6
Renal failure acute (Renal and urinary disorders) | 5
Renal failure chronic (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Swelling face (Skin and subcutaneous tissue disorders) | 1
Endotracheal intubation (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 2
Femoral artery embolism (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypertensive emergency (Vascular disorders) | 1
Hypotension (Vascular disorders) | 5
Phlebitis superficial (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=282)
Anaemia (Blood and lymphatic system disorders) | 16
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 29
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 22
Pyrexia (General disorders) | 28
Hyperkalaemia (Metabolism and nutrition disorders) | 14
Hypoglycaemia (Metabolism and nutrition disorders) | 15
Hypokalaemia (Metabolism and nutrition disorders) | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 15
Insomnia (Psychiatric disorders) | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14
Hypotension (Vascular disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.